CLINICAL TRIAL: NCT01316081
Title: A 4-month, Randomized, Placebo-controlled, Double-blind Intervention of Antioxidant Supplementation in Overweight Children Enrolled in an Outpatient Weight-loss Program: Effects on Oxidative and Inflammatory Markers, Hepcidin, Iron Status, and Components of the Metabolic Syndrome
Brief Title: A 4-month Intervention of Antioxidant Supplementation in Overweight Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, The Principal Investigator, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Aox_obesity_SM
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Metabolic Syndrome
Keywords: antioxidant supplementation; childhood obesity; hepcidin; iron status; oxidative stress; inflammation
MeSH Terms: conditions — Metabolic Syndrome; Pediatric Obesity; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Antioxidant Group (Experimental): 500mg Vitamin C 400 I.E. Vitamin E 50 mcg Selenium
  Interventions: Dietary Supplement: Vitamin C Vitamin E Selenvital all from Burgerstein Vitamine
- Placebo Group (Placebo Comparator): identical appearing placebo supplements
  Interventions: Dietary Supplement: Vitamin C Vitamin E Selenvital all from Burgerstein Vitamine

INTERVENTIONS:
Dietary Supplement: Vitamin C Vitamin E Selenvital all from Burgerstein Vitamine — Vitamin C: 500mg Vitamin E: 400 I.U. Selenium: 50mcg
  Placebo Supplements: identical appearing tablets
  Other Names: Burgerstein Vitamin C retard 500mg SWISSMEDIC Nr. 44259028; Burgerstein Vitamin E 400 I.E. SWISSMEDIC Nr. 44562014; Burgerstein Selenvital 50µg

SUMMARY:
In obese children, low antioxidant vitamin intake and reduced antioxidant capacity are common. Weight reduction reduces subclinical inflammation in obese subjects, and, similarly, antioxidant vitamins have been shown to reduce the expression of proinflammatory cytokines. Moreover, antioxidants reduce oxidative stress which influences endothelial function and might play a crucial role in the pathogenesis of obesity-related disorders. Furthermore, overweight children and adults have a markedly increased risk for iron deficiency. The mechanism linking obesity with iron deficiency is unclear. Growing evidence suggests that the elevated inflammatory status associated with obesity increases circulating hepcidin and this contributes to iron deficiency. Weight reduction has been shown to be associated with reduced inflammation and serum hepcidin concentrations, and an improved functional iron state. Thus, reducing inflammation in obese children may improve iron metabolism and reduce their risk of iron deficiency.

Therefore, positive effects on subclinical inflammation, hepcidin/iron status and metabolic risk factors in obese children during weight loss may be enhanced by supplementation with antioxidants.

The aim of the present study is to investigate the effect of 4-month antioxidant supplementation on subclinical inflammation, hepcidin, iron status and components of the metabolic syndrome in overweight children undergoing an outpatient weight-loss program.

Our hypotheses are: 1. During an outpatient weight loss program, antioxidant supplementation will reduce oxidative and inflammatory stress associated with obesity to a greater extent than weight loss alone. 2. This will have two effects, compared to weight loss alone: a.It will reduce circulating hepcidin concentrations, and improve iron status. b.It will improve metabolic and cardiovascular risk factors.

Subjects The investigators plan to enroll 50 children who are participants in outpatient weight-loss programs in the German part of Switzerland. Enrollment will be done with the agreement and assistance of the physician supervising the weight-loss program, and the timing of the study measurements will be incorporated within the existing program schedule. It is anticipated that the baseline blood sample for this study will be obtained from the regular baseline venipuncture for the weight-loss study. Criteria for participation include age between 10 to 18 years and a BMI over the 85th percentile for age and sex. Exclusion criteria include major medical illnesses, including gastrointestinal, inflammatory, bleeding and/or endocrine disorders, a history of nephrolithiasis, unusual dietary habits (e.g. vegetarianism), major food allergies or intolerances (lactose, gluten), smoking, and use of chronic medications or vitamin/mineral antioxidant supplements.

Study design The study will be a double-blind, randomized, placebo-controlled intervention trial. Children will be randomly assigned to one of two groups: antioxidant (AO) or placebo (P) supplement. If it is necessary to enroll children from different weight-loss programs, then randomization will be stratified by program. During the 4-month weight loss period, the AO group will consume oral supplements of ascorbic acid (500mg), alpha tocopherol (400 IU), and 50 µg selenium (all from Burgerstein Vitamins, Rapperswil-Jona, Switzerland) each evening with diner, whereas the P group will consume identical-appearing placebo supplements.

ELIGIBILITY:
Inclusion Criteria:

* age between 10 to 18 years old
* BMI over the 85th percentile for age and sex

Exclusion Criteria:

* history of nephrolithiasis
* history of bleeding disorder
* smoking
* type 2 diabetes
* NAFLD
* Asthma

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
oxidative markers (isoprostanes) | blood sample after 4 months
inflammatory parameters | blood sample after 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Zimmermann, Prof, Principal Investigator — ETH Zurich
Locations (1):
- Swiss Federal Institute of Technology , Laboratory of Human Nutrition, Zurich, Switzerland

REFERENCES:
- [Derived] Murer SB, Aeberli I, Braegger CP, Gittermann M, Hersberger M, Leonard SW, Taylor AW, Traber MG, Zimmermann MB. Antioxidant supplements reduced oxidative stress and stabilized liver function tests but did not reduce inflammation in a randomized controlled trial in obese children and adolescents. J Nutr. 2014 Feb;144(2):193-201. doi: 10.3945/jn.113.185561. Epub 2013 Dec 18. PMID 24353344